CLINICAL TRIAL: NCT05109234
Title: A Multicenter, Open-Label, Single-Arm Study to Evaluate Long-Term Safety, Tolerability, and Efficacy of Brivaracetam in Study Participants 2 to 26 Years of Age With Childhood Absence Epilepsy or Juvenile Absence Epilepsy
Brief Title: A Study to Test the Long-term Safety, Tolerability and Efficacy of Brivaracetam in Study Participants 2 to 26 Years of Age With Childhood Absence Epilepsy or Juvenile Absence Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0132; 2020-002769-33 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Childhood Absence Epilepsy; Juvenile Absence Epilepsy
Keywords: Childhood absence epilepsy; Juvenile absence epilepsy; Brivaracetam; Phase 3; Briviact; CAE; JAE; Epilepsy
MeSH Terms: conditions — Epilepsy, Absence; Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Brivaracetam arm (Experimental): Subjects in this arm will receive various brivaracetam doses as oral solution or film-coated tablet twice per day.
  Interventions: Drug: Brivaracetam Film-coated tablet; Drug: Brivaracetam oral solution

INTERVENTIONS:
Drug: Brivaracetam Film-coated tablet — * Pharmaceutical form: Film-coated tablet
  * Route of administration: Oral use
  Brivaracetam film-coated tablet [10, 25 or 50 mg] will be administered twice per day in equal doses.
Drug: Brivaracetam oral solution — * Pharmaceutical form: Oral solution
  * Route of administration: Oral use
  Brivaracetam oral solution [10 mg/mL]) will be administered twice per day in equal doses.

SUMMARY:
The purpose of the study is to investigate the long-term safety, tolerability and efficacy of brivaracetam in pediatric study participants with childhood absence epilepsy (CAE) or juvenile absence epilepsy (JAE).

ELIGIBILITY:
Inclusion Criteria:

* Participants who previously participated in N01269 (NCT04666610) and qualify for entry into EP0132 as per N01269 (NCT04666610) protocol with a confirmed diagnosis of childhood absence epilepsy (CAE) or juvenile absence epilepsy (JAE), and for whom a reasonable benefit from long-term administration of brivaracetam (BRV) is expected, in the opinion of the Investigator
* A sexually active male study participant must agree to use contraception during the treatment period and for at least 2 days, corresponding to the time needed to eliminate study treatment, after the last dose of study treatment and refrain from donating sperm during this period
* A female study participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

  1. The study participant is premenarchal OR
  2. A woman of childbearing potential (WOCBP) who agrees to follow the contraceptive guidance during the treatment period and for at least 2 days after the last dose of study medication, corresponding to the time needed to eliminate study treatment
* Study participant is capable of and provides consent/assent, and the study participant's parent/legal representative/caregiver provides signed informed consent for minor study participants, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

* Study participant has a history or presence of paroxysmal nonepileptic seizures
* Study participant has severe medical, neurological, or psychiatric disorders or laboratory values, which could, at the discretion of the Investigator, affect safe participation in the study or would preclude appropriate study participation
* Study participant has a clinically relevant electrocardiogram (ECG) abnormality in the opinion of the Principal Investigator
* Study participant has hepatic impairment (Child Pugh Score A, B, or C) based on the Investigator's assessment
* Study participant has active suicidal ideation prior to study entry as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia Suicide Severity Rating Scale (C-SSRS) (for study participants 6 years or older) or clinical judgment (for study participants younger than 6 years). The study participant should be referred immediately to a Mental Healthcare Professional
* Study participant has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt). The Investigator must immediately refer the study participant to a Mental Healthcare Professional
* Participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Participant has a known fructose intolerance or known hypersensitivity to any components of brivaracetam (BRV) or excipients or a drug with similar chemical structure. Note that the tablets contain lactose
* Study participant has end-stage kidney disease requiring dialysis
* Concomitant use of carbamazepine, felbamate, gabapentin, oxcarbazepine, phenobarbital, phenytoin, tiagabine, or vigabatrin
* Study participant has planned participation in any clinical study on an investigational drug or device
* Study participant has poor compliance with the visit schedule or medication intake in the core study in the opinion of the Investigator

Ages: 2 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (24):
- United States (5):
  - Ep0132 115, Birmingham, Alabama
  - Ep0132 105, Orange, California
  - Ep0132 110, Augusta, Georgia
  - Ep0132 100, New Brunswick, New Jersey
  - Ep0132 109, Winston-Salem, North Carolina
- Georgia (5):
  - Ep0132 400, Tbilisi
  - Ep0132 401, Tbilisi
  - Ep0132 402, Tbilisi
  - Ep0132 403, Tbilisi
  - Ep0132 405, Tbilisi
- Italy (6):
  - Ep0132 323, Messina
  - Ep0132 321, Milan
  - Ep0132 320, Pavia
  - Ep0132 322, Roma
  - Ep0132 325, Roma
  - Ep0132 326, Verona
- Romania (3):
  - Ep0132 562, Bucharest
  - Ep0132 560, Iași
  - Ep0132 561, Timişoara, Judeţ Timiş
- Slovakia (2):
  - Ep0132 632, Bardejov
  - Ep0132 630, Dubnica nad Váhom
- Ukraine (3):
  - Ep0132 600, Dnipro
  - Ep0132 601, Dnipro
  - Ep0132 607, Uzhhorod

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in March 2022 and concluded in March 2025.
Pre-assignment Details: The Participant Flow refers to the Safety Set (SS). Participants who participated in N01269 (NCT04666610) were offered participation in this study.
Groups:
- Childhood Absence Epilepsy (CAE): Brivaracetam: Participants with CAE entered the Evaluation Period and received a Brivaracetam (BRV) tablet or oral solution dose of 100 mg/day (or equivalent dose of 2 mg/kg/day for study participants weighing less than 50kg). The dose could be adjusted after 3 days in the range of 50 to 200 mg/day (or equivalent dose of 1 to 4 mg/kg/day for study participants weighing less than 50 kg) based on the individual needs. The maximum allowed daily dose was 200 mg/day (or equivalent dose of 4 mg/kg/day for study participants weighing less than 50 kg). The duration of the study per study participant was 2 years at minimum, until approval of BRV for the indication of CAE was obtained for pediatric participants in their age range, until a managed access program (MAP) was established as allowed per country-specific requirements in addition to legal and regulatory guidelines, or until the investigational product development in the related indication is stopped by the Sponsor, whichever come first. For study participants who transitioned to another BRV study EP0224 (NCT06315322) or a managed access program or similar type of program or who convert to commercial BRV (if, when, and where available), the final visit (FV) instead of the early discontinuation visit (EDV) needed to be completed; however, down-titration (dose reduction to half during 4 weeks) and the Safety Visit (SV) were not applicable in such a case.
- Juvenile Absence Epilepsy (JAE): Brivaracetam: Participants with JAE entered the Evaluation Period and received a Brivaracetam (BRV) tablet or oral solution dose of 100 mg/day (or equivalent dose of 2 mg/kg/day for study participants weighing less than 50 kg). The dose could be adjusted after 3 days in the range of 50 to 200 mg/day (or equivalent dose of 1 to 4 mg/kg/day for study participants weighing less than 50 kg) based on the individual needs. The maximum allowed daily dose was 200 mg/day (or equivalent dose of 4 mg/kg/day for study participants weighing less than 50 kg). The duration of the study per study participant was 2 years at minimum, until approval of BRV for the indication of JAE was obtained for pediatric participants in their age range, until a MAP was established as allowed per country-specific requirements in addition to legal and regulatory guidelines, or until the investigational product development in the related indication is stopped by the Sponsor, whichever come first. For study participants who transitioned to another BRV study EP0224 (NCT06315322) or a managed access program or similar type of program or who convert to commercial BRV (if, when, and where available), the FV instead of the EDV needed to be completed; however, down-titration (dose reduction to half during 4 weeks) and the SV were not applicable in such a case.
Period: Overall Study
Arm/Group | Childhood Absence Epilepsy (CAE): Brivaracetam | Juvenile Absence Epilepsy (JAE): Brivaracetam
Started | 64 | 20
Evaluation Period (Up to 24 Months) (Participants who were enrolled in the study will enter the Evaluation Period and received the BRV dose.) | 64 | 20
Completed | 50 | 14
Not Completed | 14 | 6
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 5 | 0
Not completed — Consent withdrawn by Participant (not due to AE) | 1 | 0
Not completed — Consent withdrawn by parent/guardian (not AE) | 3 | 4
Not completed — Evacuated from Ukraine due to the war | 2 | 0
Not completed — Missed safety visit; study incomplete per protocol | 1 | 0

BASELINE CHARACTERISTICS:
Population: The SS consisted of all enrolled study participants who took at least 1 dose of study drug in the long-term follow-up (LTFU) study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Childhood Absence Epilepsy (CAE): Brivaracetam | Juvenile Absence Epilepsy (JAE): Brivaracetam | Total
Number analyzed (Participants) | 64 | 20 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.56 (2.49) | 13.93 (1.64) | 10.60 (2.97)
Age, Customized [Count of Participants; unit: Participants]
  24 months - <12 years | 53 | 2 | 55
  12 - <18 years | 11 | 18 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 11 | 48
  Male | 27 | 9 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 0 | 1
  Race: Black or African American | 5 | 0 | 5
  Race: White | 57 | 20 | 77
  Race: Other or Mixed | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 5 | 0 | 5
  Ethnicity: Not Hispanic or Latino | 59 | 20 | 79

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. TEAEs are defined as AEs that had onset on or after the day of first dose of BRV.
Time Frame: From Entry Visit up to 16.32 months (median); min, max exposure to BRV was (0.4, 31.0) months
Population: The SS consisted of all enrolled study participants who took at least 1 dose of study drug in the LTFU study.
Measure: Number; unit: percentage of participants
Arm/Group | Childhood Absence Epilepsy (CAE): Brivaracetam | Juvenile Absence Epilepsy (JAE): Brivaracetam
Number analyzed (Participants) | 64 | 20
percentage of participants | 42.2 | 55.0

2. Primary Outcome: Percentage of Participants With TEAEs Leading to Discontinuation of Study Treatment
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. TEAEs are defined as AEs that had onset on or after the day of first dose of BRV. Percentage of participants with TEAEs leading to discontinuation were reported.
Time Frame: From Entry Visit up to 16.32 months (median); min, max exposure to BRV was (0.4, 31.0) months
Population: The SS consisted of all enrolled study participants who took at least 1 dose of study drug in the LTFU study.
Measure: Number; unit: percentage of participants
Arm/Group | Childhood Absence Epilepsy (CAE): Brivaracetam | Juvenile Absence Epilepsy (JAE): Brivaracetam
Number analyzed (Participants) | 64 | 20
percentage of participants | 3.1 | 10.0

3. Secondary Outcome: Percentage of Participants With Serious TEAEs
Description: TEAEs are defined as AEs that had onset on or after the day of first dose of BRV. A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires in patient hospitalization or prolongation of existing hospitalization, is a congenital anomaly or birth defect, results in permanent or significant disability/incapacity, other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Entry Visit up to 16.32 months (median); min, max exposure to BRV was (0.4, 31.0) months
Population: The SS consisted of all enrolled study participants who took at least 1 dose of study drug in the LTFU study.
Measure: Number; unit: percentage of participants
Arm/Group | Childhood Absence Epilepsy (CAE): Brivaracetam | Juvenile Absence Epilepsy (JAE): Brivaracetam
Number analyzed (Participants) | 64 | 20
percentage of participants | 3.1 | 10.0

4. Secondary Outcome: Percentage of Participants With Study Drug-related TEAEs
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. TEAEs are defined as AEs that had onset on or after the day of first dose of BRV. Drug related AEs are the subset of AEs that the investigator considers as related to the study drug.
Time Frame: From Entry Visit up to 16.32 months (median); min, max exposure to BRV was (0.4, 31.0) months
Population: The SS consisted of all enrolled study participants who took at least 1 dose of study drug in the LTFU study.
Measure: Number; unit: percentage of participants
Arm/Group | Childhood Absence Epilepsy (CAE): Brivaracetam | Juvenile Absence Epilepsy (JAE): Brivaracetam
Number analyzed (Participants) | 64 | 20
percentage of participants | 6.3 | 10.0

5. Secondary Outcome: Percentage of Participants With Absence Seizure Freedom Within 4 Days Prior to or During the 1-hour Electroencephalogram (EEG)
Description: A 1-hour EEG was performed. The awake hours from the EEG was analyzed for absence seizures. Every 1-hour EEG included hyperventilation as a standard provocation test at the beginning of the EEG. Participant was regarded as not meeting the criteria for absence seizure freedom if they received any permitted antiepileptic drugs including benzodiazepine in the 4 days prior to the EEG or during the EEG. Participants who continue in the study beyond 2 years have their data truncated at Year 2 Month 24 yearly evaluation visit (YEV).
Time Frame: Full Evaluation Visit (6 months), Yearly Evaluation Visit (12 months), Full Evaluation Visit (18 months), Yearly Evaluation Visit (24 months)
Population: The SS consisted of all enrolled study participants who took at least 1 dose of study drug in the LTFU study. Here, overall number of participants analyzed included all participants who were evaluable for this assessment and number analyzed (n) signifies participants who were evaluable at each specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Childhood Absence Epilepsy (CAE): Brivaracetam | Juvenile Absence Epilepsy (JAE): Brivaracetam
Number analyzed (Participants) | 56 | 20
percentage of participants
  FEV: 6 months | 46.4 | 70.0
  YEV: 12 months: number analyzed (Participants) | 47 | 18
  YEV: 12 months | 42.6 | 44.4
  FEV: 18 months: number analyzed (Participants) | 36 | 16
  FEV: 18 months | 38.9 | 50.0
  YEV: 24 months: number analyzed (Participants) | 30 | 11
  YEV: 24 months | 26.7 | 18.2

6. Secondary Outcome: Percentage of Participants With Absence Seizure Freedom Based on Daily Seizure Diary Over the Entire Evaluation Period and by 3-month Time Intervals
Description: During the study, participants kept a diary to record daily seizure activity from entry visit (Visit 1) until the final visit. Each seizure type experienced were recorded. The participant was considered as not meeting the criteria for absence seizure freedom if they use any permitted anti-epileptic drugs at anytime during the period, and/or complete less than 80% of diaries during the period. Evaluation Period includes all daily seizure diary data over the Evaluation Period up to Month 24 YEV, this includes data from the end of Months 22 to 24 up to the Month 24 YEV where this data is truncated. If a participant does not attend the Month 24 YEV then data was truncated at the last day the participant is in the Evaluation Period in the Month 24 YEV window. Participants who continue in the study beyond 2 years have their data truncated at Year 2 Month 24 YEV, or the last day the participant was in the Evaluation Period in the Month 24 YEV window if this visit is not attended.
Time Frame: Months 1-3, Months 4-6, Months 7-9, Months 10-12, Months 13-15, Months 16-18, Months 19-21, Months 22-24 and Entire Evaluation Period (Up to 24 months)
Population: The SS consisted of all enrolled study participants who took at least 1 dose of study drug in the LTFU study. Here, "n" signifies participants who were evaluable at each specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Childhood Absence Epilepsy (CAE): Brivaracetam | Juvenile Absence Epilepsy (JAE): Brivaracetam
Number analyzed (Participants) | 64 | 20
percentage of participants
  Months 1-3 | 34.4 | 35.0
  Months 4-6: number analyzed (Participants) | 59 | 20
  Months 4-6 | 39.0 | 55.0
  Months 7-9: number analyzed (Participants) | 53 | 19
  Months 7-9 | 37.7 | 57.9
  Months 10-12: number analyzed (Participants) | 49 | 18
  Months 10-12 | 38.8 | 55.6
  Months 13-15: number analyzed (Participants) | 44 | 18
  Months 13-15 | 31.8 | 61.1
  Months 16-18: number analyzed (Participants) | 39 | 16
  Months 16-18 | 35.9 | 56.3
  Months 19-21: number analyzed (Participants) | 33 | 14
  Months 19-21 | 30.3 | 42.9
  Months 22-24: number analyzed (Participants) | 32 | 12
  Months 22-24 | 21.9 | 33.3
  Entire Evaluation Period (up to 24 months) | 28.1 | 30.0

ADVERSE EVENTS:
Time Frame: From Entry Visit up to 16.32 months (median); min, max exposure to BRV was (0.4, 31.0) months
Description: Treatment-emergent adverse events were defined as AEs that had onset on or after the day of first dose of BRV. The Safety Set (SS) consisted of all enrolled study participants who took at least 1 dose of study drug in the LTFU study.
Arm/Group | Childhood Absence Epilepsy (CAE): Brivaracetam | Juvenile Absence Epilepsy (JAE): Brivaracetam
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/64 | 2/20
Other Adverse Events (participants affected / at risk) | 15/64 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Childhood Absence Epilepsy (CAE): Brivaracetam (N=64) | Juvenile Absence Epilepsy (JAE): Brivaracetam (N=20)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Measles (Infections and infestations) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Childhood Absence Epilepsy (CAE): Brivaracetam (N=64) | Juvenile Absence Epilepsy (JAE): Brivaracetam (N=20)
Pyrexia (General disorders) | 4 (4) | 4 (5)
Petit mal epilepsy (Nervous system disorders) | 9 (10) | 5 (8)
Headache (Nervous system disorders) | 3 (4) | 2 (3)

LIMITATIONS AND CAVEATS:
EP0132 enrolled fewer participants than expected (approximately 140) so it was closed prematurely, followed by the initiation of the managed access program EP0225 (NCTID not applicable) and its replacement with the new open-label study EP0224 (NCT06315322).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT05109234/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT05109234/SAP_001.pdf